CLINICAL TRIAL: NCT00205153
Title: A Team Model of Hypertension Care in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-2000-0284; NIH R01 HL78580
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension
Keywords: hypertension in African Americans
MeSH Terms: conditions — Hypertension | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEAM Care (Experimental): Intervention pharmacies implement 6-month TEAM program.
  Interventions: Behavioral: Pharmacy TEAM monitoring and counseling
- Usual Care (No Intervention): Control pharmacies provide "usual care" only.

INTERVENTIONS:
Behavioral: Pharmacy TEAM monitoring and counseling — Pharmacy team monitors and counsels patient using automatic BP monitors and special TEAM tools for assessing and improving patient adherence, barriers to adherence, lifestyle, drug therapy, BP control, and collaboration with physicians.
  Arms: TEAM Care

SUMMARY:
This Team Education and Adherence Monitoring (TEAM) trial will evaluate the cost-effectiveness of a pharmacy-based intervention in a randomized controlled trial involving 597 treated hypertensive African American patients in five Wisconsin cities. The study involves 28 community pharmacies (14 intervention, 14 control) owned by two pharmacy corporations. Intervention pharmacists and pharmacy technicians implemented a 6-month blood pressure (BP) monitoring program that involved working together as a team with patients and their physicians to achieve improved medication adherence, healthy lifestyles, drug therapy, and hypertension control.

DETAILED DESCRIPTION:
Researchers screened and enrolled 20-25 subjects in each study pharmacy. Intervention pharmacists and technicians attended a 7-hour TEAM training program on BP monitoring, JNC 7 guidelines, and specially designed tools for assessing and improving medication adherence, lifestyle, patient scheduling and retention, and collaboration with physicians. Intervention teams received specially designed tools, automatic BP monitors, and furniture for setting up and implementing a blood pressure clinic at their pharmacy. Staff from control pharmacies received printed information only and provided "usual care". Outcomes will be determined by blinded data collectors who will re-check patients' BPs and administer follow-up surveys after 6 and 12 months. Researchers also will survey pharmacy staff and review pharmacy records to determine changes in refill adherence and prescribing.

ELIGIBILITY:
Inclusion Criteria:is African American and 18 years old or older; has active prescription for BP drug; obtains all BP drugs at the study pharmacy; is able to read and fill out short questionnaires; is able to come to pharmacy for 6 monthly pharmacy visits if needed; has screening BP between 140/90 mm Hg and 210/115 mm Hg.

Exclusion Criteria: history of organ transplant or kidney dialysis, symptoms of advanced congestive heart failure, memory impairment that interferes with daily functioning,terminal illness,pregnancy, alcohol or substance abuse problem,physician recommendation of exclusion for other condition that may require special care or limit participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving hypertension control | 6 months after enrollment
change in systolic and diastolic blood pressure | 6 months after enrollment

SECONDARY OUTCOMES:
patient adherence to drug regimen | 6 months after enrollment
pharmacist adherence to TEAM protocol (intervention fidelity) | 6 months after enrollment
change in drug prescribing | 6 months after enrollment
patient-reported barriers to adherence (e.g. bothersome side effects) | 6 months after enrollment
cost-effectiveness of pharmacy intervention | 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie L Svarstad, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin School of Pharmacy, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Svarstad BL, Brown RL, Shireman TI. A successful intervention to improve medication adherence in Black patients with hypertension: Mediation analysis of 28-site TEAM trial. J Am Pharm Assoc (2003). 2022 May-Jun;62(3):800-808.e3. doi: 10.1016/j.japh.2022.01.002. Epub 2022 Jan 6. PMID 35120864
- [Derived] Shireman TI, Svarstad BL. Cost-effectiveness of Wisconsin TEAM model for improving adherence and hypertension control in black patients. J Am Pharm Assoc (2003). 2016 Jul-Aug;56(4):389-96. doi: 10.1016/j.japh.2016.03.002. Epub 2016 May 13. PMID 27184784
- [Derived] Svarstad BL, Kotchen JM, Shireman TI, Brown RL, Crawford SY, Mount JK, Palmer PA, Vivian EM, Wilson DA. Improving refill adherence and hypertension control in black patients: Wisconsin TEAM trial. J Am Pharm Assoc (2003). 2013 Sep-Oct;53(5):520-9. doi: 10.1331/JAPhA.2013.12246. PMID 24030130